CLINICAL TRIAL: NCT01013220
Title: Influencing Employer Purchasing Behavior
Brief Title: Depression Management at the Workplace
Acronym: DMW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Colorado Business Group on Health (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH076227 (NIH)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: depression; depression care management; financing; absenteeism; presenteeism; employer decisions to purchase health care benefits
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depression Product Detailing (Experimental): Employers receive education on how to purchase high quality depression management products to improve the quality of depression treatment depressed employees receive. Materials delivered in this arm of the study are available at www.caremanagementfordepression.org
  Interventions: Other: Depression Product Detailing
- Depression HEDIS Detailing (Placebo Comparator): Employers receive education on how to obtain and use HEDIS depression indicators to encourage health plans to improve the quality of depression treatment depressed employees receive
  Interventions: Other: Depression HEDIS detailing

INTERVENTIONS:
Other: Depression Product Detailing — 1. two hour academic detailing of depression management products to employees with responsibility for purchasing health care benefits
  2. technical assistance in purchasing high quality depression management products
  Arms: Depression Product Detailing
Other: Depression HEDIS detailing — 1. academic detailing to employees responsible for purchasing health care benefits on how to use HEDIS indicators for depression to assure their depressed employees receive high quality care for the condition
  2. technical assistance
  Arms: Depression HEDIS Detailing

SUMMARY:
Randomized trials demonstrate that depression management products can improve clinical and organizational outcomes sufficiently for selected employers to realize a return on investment. Rather than usual care marketing which uses voltage-enhanced promises to sell voltage-diminished products, the investigators designed an evidence-based (EB) intervention to encourage employers to purchase a depression management product that offers the type, intensity and duration of care shown to provide clinical and organizational value. In an RCT designed to examine employer benefit purchasing behavior of depression products in 360 employer members of over 20 regional business coalitions, the research team proposes: (a) to compare the impact of evidence-based (EB) to usual care (UC) presentations on employer benefit purchasing behavior, and (b) to identify mediators and organizational moderators of intervention impact on employer benefit purchasing behavior.

This study addresses what policy analysts argue is one of the most pivotal problems in the translation of evidence-based care to 'real world' settings: whether purchasers can be influenced to buy health care products on the basis of value rather than cost. In the likely event that EB > UC, the study will provide encouragement to use an evidence-based approach to market new health care products to private payers on the basis of the product's clinical and organizational value. UC may achieve comparable outcomes to EB if the limiting factors in benefit purchasing are organizational, purchasing group and vendor constraints that no intervention can meaningfully modify. Support for this scenario would encourage the targeted marketing of new products to coalition members with empirically identified organizational, purchasing group and vendor characteristics, using usual care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Coalitions who belong to the National Business Coalition on Health are eligible if:

  * they have 30+ employer purchasers/affiliates as members
  * they act as more than purchasing agents
  * (3)they did not participate in the research team's preliminary studies on this topic.
* Employers of participating coalitions are eligible if:

  * they are a public or private organization providing health care benefits to 100+ domestic employees
  * they have not purchased a depression management product in the past two years.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
employer purchase of depression management product | two years after intervention

SECONDARY OUTCOMES:
fidelity of depression management model purchased to evidence-based models | two years after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Rost, PhD, Principal Investigator — Florida State University, College of Medicine
Locations (1):
- Colorado Business Group on Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Rost KM, Meng H, Xu S. Work productivity loss from depression: evidence from an employer survey. BMC Health Serv Res. 2014 Dec 18;14:597. doi: 10.1186/s12913-014-0597-y. PMID 25519705
- [Derived] Rost KM, Marshall D, Xu S. Intervention impact on depression product appraisal and purchasing behavior by employers: a randomized trial. BMC Health Serv Res. 2014 Sep 24;14:426. doi: 10.1186/1472-6963-14-426. PMID 25248854
- See also: materials for academic detailing of depression management products — http://www.caremanagementfordepression.org